CLINICAL TRIAL: NCT00693121
Title: Amantadine Hydrochloride for Treatment of Symptoms of the Post-traumatic Confusional State Among Neurorehabilitation Admissions With TBI: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Amantadine for Treatment of Symptoms of the Post-traumatic Confusional State
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Methodist Rehabilitation Center (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Theresa San Augustin, National Institute for Disability and Rehabilitation Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MethodistRC Project 1; NIDRR grant #: H133A020514
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2008-06

CONDITIONS: Traumatic Brain Injury; Posttraumatic Confusional State; Delirium
Keywords: Traumatic Brain Injury; Posttraumatic Confusional State; Delirium; Amantadine; Clinical trial
MeSH Terms: conditions — Brain Injuries, Traumatic; Delirium | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Identical capsule to amantadine hydrochloride active intervention, administered twice daily x 14 days
  Interventions: Drug: Placebo capsule
- Amantadine (Active Comparator): Amantadine hydrochloride 100mg capsule administered twice daily x 14 days
  Interventions: Drug: Amantadine hydrochloride

INTERVENTIONS:
Drug: Amantadine hydrochloride — 100mg administered orally twice daily x 14 days
  Arms: Amantadine
Drug: Placebo capsule — capsule, identical to amantadine hydrochloride capsule, administered twice daily x 14 days
  Arms: Placebo

SUMMARY:
Patients with traumatic brain injury often experience a period of acute confusion that may include agitation as they recover from their injuries. While this confusion generally resolves with time, patients may pose increased risk of injury to themselves or others during this period. Their behavior may also increase stress for family members and interfere with their ability to benefit from rehabilitation therapies. A number of different medications have been used to treat confusion to decrease agitation, decrease risk of injury, and improve participation in rehabilitation therapies. To this point, there has not been a research or scientific basis for knowing which medication is the best for a specific patient. The overall goal of this study is to conduct a scientific investigation to help determine which medication works best to treat confusion.

Study hypothesis: Amantadine will reduce the severity and number of symptoms of acute confusion after traumatic brain injury.

DETAILED DESCRIPTION:
Patients with TBI who require inpatient rehabilitation are frequently confused at the time of admission for rehabilitation. Our investigations of confusion conducted as part of the TBIMSM have clarified the nature of confusion in early recovery after TBI. Early confusion (PTCS) has been found to be a complex syndrome characterized by disorientation, cognitive impairment, restlessness, decreased level of daytime arousal, sleep disturbance, fluctuation of symptoms, and psychotic-type symptoms. PTCS complicates early management of patients with TBI, and may contribute to increased risk of injury to patients and hospital staff, increased stress among family members and staff, decreased participation in therapies, increased cost of care, and an increased likelihood of being discharged to psychiatric or long-term care settings. These facts indicate the need for effective management of PTCS. Consensus regarding optimal treatment of the cognitive and behavioral symptoms encountered among patients with PTCS does not exist currently. While many agents have been tried to address such symptoms in TBI, few have been investigated systematically. These circumstances indicate the need for appropriate clinical trials to provide guidance to clinicians for medical treatment of PTCS. In response, the NIDRR-Traumatic Brain Injury Model System of Mississippi proposed a randomized, double-blinded, placebo-controlled, parallel group trial for the pharmacological treatment of PTCS. The agent selected for this clinical trial is amantadine, an NMDA and indirect dopamine agonist. This agent will be compared to placebo on response measures of efficacy and safety.

Study hypothesis: Amantadine will reduce the severity and number of symptoms of PTCS.

ELIGIBILITY:
Inclusion Criteria:

* Acute Traumatic Brain Injury (≤90 days postinjury)
* Responsive (not fulfilling criteria for Minimally Conscious State)
* Meet PTCS criteria on 2 consecutive examinations (as determined by the Confusion Assessment Protocol)
* Initial neurorehabilitation hospital admission
* Anticipated ≥2 week length-of-stay after meeting PTCS criteria

Exclusion Criteria:

* Preexisting seizure disorder
* Prior history of hospitalization for psychiatric condition

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-04; Primary Completion 2007-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Confusion Assessment Protocol (number of symptoms) | 14 days

SECONDARY OUTCOMES:
number of participants withdrawn from study due to fulfillment of "escape criteria" | 14 days
Time to reach "non-confused" Confusion Assessment Protocol score | <14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Yablon, M.D., Principal Investigator — Brain Injury Program, Methodist Rehabilitation Center; Mark Sherer, Ph.D., Study Director — Department of Research, Memorial Hermann/TIRR, Houston, TX; Risa N Richardson, Ph.D., Study Director — Polytrauma Program, James A. Haley Veterans Hospital, Tampa, FL
Locations (1):
- Methodist Rehabilitation Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Sherer M, Yablon SA, Nakase-Richardson R, Nick TG. Effect of severity of post-traumatic confusion and its constituent symptoms on outcome after traumatic brain injury. Arch Phys Med Rehabil. 2008 Jan;89(1):42-7. doi: 10.1016/j.apmr.2007.08.128. PMID 18164329
- [Background] Nakase-Richardson R, Yablon SA, Sherer M. Prospective comparison of acute confusion severity with duration of post-traumatic amnesia in predicting employment outcome after traumatic brain injury. J Neurol Neurosurg Psychiatry. 2007 Aug;78(8):872-6. doi: 10.1136/jnnp.2006.104190. Epub 2006 Dec 18. PMID 17178822
- [Background] Sherer M, Nakase-Thompson R, Yablon SA, Gontkovsky ST. Multidimensional assessment of acute confusion after traumatic brain injury. Arch Phys Med Rehabil. 2005 May;86(5):896-904. doi: 10.1016/j.apmr.2004.09.029. PMID 15895334
- [Background] Nakase-Thompson R, Sherer M, Yablon SA, Nick TG, Trzepacz PT. Acute confusion following traumatic brain injury. Brain Inj. 2004 Feb;18(2):131-42. doi: 10.1080/0269905031000149542. PMID 14660226